CLINICAL TRIAL: NCT02760888
Title: Oral Tramadol Versus Diclofenac For Pain Relief Before Outpatient Hysteroscopy: A Randomized Controlled Trial
Brief Title: Oral Tramadol Versus Diclofenac For Pain Relief Before Outpatient Hysteroscopy:
Acronym: OPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Assistant professor of Obstetrics and Gynecology Faculty of Medicine Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EDCU HY
Record Dates: First submitted 2016-04-30; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2015-12

CONDITIONS: Pain, Procedure
MeSH Terms: conditions — Pain | interventions — Tramadol; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Tramadol (Active Comparator): Women will receive oral tramadol 100 mg 1 hour before the procedure
  Interventions: Drug: Tramadol
- Diclofenac (Active Comparator): Women will receive 100 mg diclofenac 1 hour before the procedure
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator): Women will receive a placebo 1 hour before the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Women will receive a oral Tramadol 100mg 1 hour before the procedure
  Arms: Tramadol
Drug: Diclofenac — Women will receive oral Diclofenac 100mg 1 hour before the procedure
  Arms: Diclofenac
Drug: Placebo — Women will receive a Placebo 1 hour before the procedure
  Arms: Placebo

SUMMARY:
The purpose of this study is there difference between the effect of Tramadol orally and Diclofenac orally with respect to : analgesic efficacy during diagnostic hysteroscopy in nulliparous women.

DETAILED DESCRIPTION:
This prospective double-blind, randomized, clinical trial, will be conducted at Ain Shams University Maternity Hospital- Early Cancer Detection Unite [ECDU].

Patients fulfilling inclusion and exclusion criteria will be divided into three groups.

Group A (study group) Include 34 patients who will receive Tramadol 100mg orally 1 hour before the procedure.

Group B (study group) Include 34 patients who will receive Diclofenac 100mg orally 1 hour before the procedure.

Group C (control group) Include 34 patients who will receive a placebo.

Pain will evaluate on two separate occasion: immediately after the procedure and 15 minutes after procedure using a 100mm line visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* BMI raging between (18.5 - 30 ).
* Scheduled for diagnostic hysteroscopy only.
* All of them should have given informed written consent.

Exclusion Criteria:

* Any contraindication to hysteroscopy (e.g. suspected pregnancy, genital tract infection).
* Receiving any other form of analgesia.
* Patients with known cervical stenosis, polyps and ulcers.
* Previous cervical surgery.
* Patients who are planning to have invasive intrauterine therapeutic interventions during the hysteroscopy.
* known sensitivity to non-steroidal anti-inflammatory and opioids drugs.
* Known gastritis or peptic ulcer or cardiac disease or Respiratory dysfunction.
* Unwilling to comply with the protocol, and Participation in another clinical trial in the last three months prior to the start of this study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Pain during the procedure | intraoperative
  Pain will be assessed using a visual analogue scale immediatly after inserting the hysterscopy
pain after the procedure | 15 minutes after completing the procedure
  15 minutes after procedure using a 100mm line visual analog scale

SECONDARY OUTCOMES:
Adverse effect and difficulties | 24 hours
  Recorded in Case Record Form

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt